CLINICAL TRIAL: NCT06157320
Title: Improving Microcirculation and Microvascular Leakage in Sepsis Patients: A Comprehensive Clinical Study of Shenfu Injection
Brief Title: Clinical Research on Shenfu Injection in Septic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 320.6750.2022-2-35
Record Dates: First submitted 2023-07-19; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-01

CONDITIONS: Sepsis
Keywords: sepsis; microcirculation; Shenfu Injection
MeSH Terms: conditions — Sepsis | interventions — Shen-Fu; Medicine, Chinese Traditional; Norepinephrine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shenfu Injection group (Experimental): within 24 hours after the diagnosis of sepsis, Shenfu injection 100 ml/day, intravenous use, continuous application for 7 days.
  Interventions: Drug: Shen-Fu
- Control group (Placebo Comparator): sepsis was treated with standardized western medicine methods
  Interventions: Drug: Norepinephrine (NE)，antibiotics，fluid resuscitation

INTERVENTIONS:
Drug: Shen-Fu — Within 24 hours of sepsis diagnosis, patients received a daily intravenous infusion of 100 ml of Shenfu Injection for a continuous duration of 7 days.
  Other Names: Traditional Chinese medicine
  Arms: Shenfu Injection group
Drug: Norepinephrine (NE)，antibiotics，fluid resuscitation — empirical antimicrobial treatment (which is promptly administered after microbial tests), fluid (crystalloids) replacement (to be established according to fluid tolerance and fluid responsiveness), and vasoactive agents (e.g., norepinephrine (NE)), which are employed to maintain mean arterial pressure above 65 mmHg and reduce the risk of fluid overload
  Other Names: Strandard treatment
  Arms: Control group

SUMMARY:
Sepsis, characterized by organ dysfunction caused by infection, exhibits increasing incidence and mortality rates, posing a significant challenge to intensive care units. Early-stage sepsis involves hemodynamic disturbances, and severe and complex microcirculatory impairments can result in tissue hypoxia and accelerate organ dysfunction. Modern medical research has indicated that the effective and rapid restoration of microcirculatory function, along with the correction of microcirculatory disorders, is a crucial aspect in the treatment of sepsis. Current guidelines recommend the use of vasoactive drugs to address hemodynamic disturbances, but their administration may further damage the microcirculation. Additionally, in patients with severe sepsis, there often exists a disparity between macrocirculatory and microcirculatory hemodynamics, and conventional clinical indicators fail to directly reflect the level of microcirculatory perfusion.

Chinese guidelines have incorporated the use of traditional Chinese medicine (TCM) in the diagnosis and treatment of sepsis, offering a new therapeutic approach to ameliorate microcirculatory impairments. This study aims to include patients with sepsis and administer Shenfu Injection via intravenous therapy. Tongue microcirculation assessment will be employed to evaluate changes in microvascular health scores, while transcutaneous oxygen and carbon dioxide pressure alterations, as well as serum lactate level variations, will be monitored to ascertain the effects of Shenfu Injection on improving early-stage microcirculatory impairments and microvascular leakage in sepsis patients. This research will clarify the clinical efficacy of Shenfu Injection in sepsis patients with microcirculatory impairments, provide evidence-based medicine and clinical evidence for TCM treatment of sepsis, and offer a solid foundation for refining sepsis treatment strategies with distinct Chinese characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Signed informed consent form;
* Meets sepsis 3.0 diagnostic criteria;

Exclusion Criteria:

* Age < 18 years;
* Known pregnancy;
* Inability to accept and complete signed informed consent within 24 hours of diagnosis of sepsis;
* Status of tracheal intubation;
* oral mucosal inflammation or damage;
* Patients with contraindications to transcutaneous oxygen partial pressure testing such as severe edema and burns;
* Concurrent participation in other treatment studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
HR:heart rate | Day0，Day1，Day 3，Day 7
  heart rate
BP:Blood pressure | Day0，Day1，Day 3，Day 7
  Blood pressure
Proportion of perfused vessels | Day0，Day1，Day 3，Day 7
  Grid-based score (3 horizontal and vertical equidistant lines). Percentage of perfused vessels per total number of vessel crossings
Microvascular fow index | Day0，Day1，Day 3，Day 7
  fow, 1 = intermittent fow, 2 = sluggish fow, 3 = normal fow Semi-quantitative assessment of the average red blood cell velocity per quadrant
Heterogeneity index | Day0，Day1，Day 3，Day 7
  Determinant of heterogeneity of blood fow, characteristic of distributive abnormalities
Hemodynamic parameters1 | Day0，Day1，Day 3，Day 7
  CI: Cardio index
Hemodynamic parameters2 | Day0，Day1，Day 3，Day 7
  SVRI:systemic vascular resistance index
Hemodynamic parameters3 | Day0，Day1，Day 3，Day 7
  GEDVI:global end-diastolic volume index

SECONDARY OUTCOMES:
Ang2:Endothelial cell function indicators | Day0，Day1，Day 3，Day 7
  Endothelial cell function indicators got from the blood of patients
VCAM1:Endothelial cell function indicators | Day0，Day1，Day 3，Day 7
  Endothelial cell function indicators got from the blood of patients
Sydecan-1:Endothelial cell function indicators | Day0，Day1，Day 3，Day 7
  Endothelial cell function indicators got from the blood of patients
6-Keto-PGF-1:Endothelial cell function indicators | Day0，Day1，Day 3，Day 7
  Endothelial cell function indicators got from the blood of patients
TXB2:Endothelial cell function indicators | Day0，Day1，Day 3，Day 7
  Endothelial cell function indicators got from the blood of patients
NO:Endothelial cell function indicators | Day0，Day1，Day 3，Day 7
  Endothelial cell function indicators got from the blood of patients
Lab test1 | Day0，Day1，Day 3，Day 7
  PH
Lab test2 | Day0，Day1，Day 3，Day 7
  PaO2 mmHg,
Lab test3 | Day0，Day1，Day 3，Day 7
  PaCO2 mmHg
Lab test4 | Day0，Day1，Day 3，Day 7
  Serum lactate mmol/L
Lab test5 | Day0，Day1，Day 3，Day 7
  IL-10 ng/ml
Lab test6 | Day0，Day1，Day 3，Day 7
  WBC ×109/L
Lab test7 | Day0，Day1，Day 3，Day 7
  Neu ×109/L
Lab test8 | Day0，Day1，Day 3，Day 7
  Lym×109/L,
Lab test9 | Day0，Day1，Day 3，Day 7
  Hb g/L,
Lab test10 | Day0，Day1，Day 3，Day 7
  PLT×109/L
Lab test11 | Day0，Day1，Day 3，Day 7
  Total bilirubin IU/L
Lab test12 | Day0，Day1，Day 3，Day 7
  Cr μmol/L
Lab test13 | Day0，Day1，Day 3，Day 7
  IL-1βng/ml
Lab test14 | Day0，Day1，Day 3，Day 7
  APTT s
Lab test15 | Day0，Day1，Day 3，Day 7
  D-Dimermg/L
Lab test16 | Day0，Day1，Day 3，Day 7
  CRP mg/L
Lab test17 | Day0，Day1，Day 3，Day 7
  ProBNP pg/ml
Lab test18 | Day0，Day1，Day 3，Day 7
  PCT ng/ml
Lab test19 | Day0，Day1，Day 3，Day 7
  TNFαng/ml
Lab test20 | Day0，Day1，Day 3，Day 7
  IL-6 ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Hongping Qu, Study Director — Shanghai Jiao Tong University Medical School Affiliated Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Gutterman DD, Chabowski DS, Kadlec AO, Durand MJ, Freed JK, Ait-Aissa K, Beyer AM. The Human Microcirculation: Regulation of Flow and Beyond. Circ Res. 2016 Jan 8;118(1):157-72. doi: 10.1161/CIRCRESAHA.115.305364. PMID 26837746
- [Result] Tian R, Wang X, Pan T, Li R, Wang J, Liu Z, Chen E, Mao E, Tan R, Chen Y, Liu J, Qu H. Plasma PTX3, MCP1 and Ang2 are early biomarkers to evaluate the severity of sepsis and septic shock. Scand J Immunol. 2019 Dec;90(6):e12823. doi: 10.1111/sji.12823. Epub 2019 Oct 7. PMID 31489646
- [Result] Tian R, Li R, Liu Y, Liu J, Pan T, Zhang R, Liu B, Chen E, Tang Y, Qu H. Metformin ameliorates endotoxemia-induced endothelial pro-inflammatory responses via AMPK-dependent mediation of HDAC5 and KLF2. Biochim Biophys Acta Mol Basis Dis. 2019 Jun 1;1865(6):1701-1712. doi: 10.1016/j.bbadis.2019.04.009. Epub 2019 Apr 16. PMID 31002870
- [Result] Yao B, Liu DW, Chai WZ, Wang XT, Zhang HM. Microcirculation dysfunction in endotoxic shock rabbits is associated with impaired S-nitrosohemoglobin-mediated nitric oxide release from red blood cells: a preliminary study. Intensive Care Med Exp. 2019 Jan 7;7(1):1. doi: 10.1186/s40635-018-0215-0. PMID 30617929
- [Result] Otero RM, Nguyen HB, Huang DT, Gaieski DF, Goyal M, Gunnerson KJ, Trzeciak S, Sherwin R, Holthaus CV, Osborn T, Rivers EP. Early goal-directed therapy in severe sepsis and septic shock revisited: concepts, controversies, and contemporary findings. Chest. 2006 Nov;130(5):1579-95. doi: 10.1378/chest.130.5.1579. PMID 17099041
- [Result] Fan KL, Wang JH, Kong L, Zhang FH, Hao H, Zhao H, Tian ZY, Yin MX, Fang H, Yang HH, Liu Y. Effect of Shen-Fu Injection () on Hemodynamics in Early Volume Resuscitation Treated Septic Shock Patients. Chin J Integr Med. 2019 Jan;25(1):59-63. doi: 10.1007/s11655-017-2965-z. Epub 2017 Oct 6. PMID 28986814
- [Result] Zhang XJ, Song L, Zhou ZG, Wang XM. Effect of shenfu injection on gastrointestinal microcirculation in rabbits after myocardial ischemia-reperfusion injury. World J Gastroenterol. 2006 Jul 21;12(27):4389-91. doi: 10.3748/wjg.v12.i27.4389. PMID 16865783
- [Result] Zhang X, Guo T, Zhang K, Guo W, An X, Gao P. Effect of shenfu injection on microcirculation in shock patients: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 Oct 23;99(43):e22872. doi: 10.1097/MD.0000000000022872. PMID 33120828
- [Result] Ince C. Hemodynamic coherence and the rationale for monitoring the microcirculation. Crit Care. 2015;19 Suppl 3(Suppl 3):S8. doi: 10.1186/cc14726. Epub 2015 Dec 18. PMID 26729241